CLINICAL TRIAL: NCT06163261
Title: Individualized and Person-centred Physical Activity and Exercise for Patients With Non Functioning Pituitary Adenoma - A Randomized Controlled Trial
Brief Title: Individualized Physical Activity or Patients With Non Functioning Pituitary Adenoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEPP
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-03

CONDITIONS: Non-functioning Pituitary Adenoma
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): This group will receive an individualized and person-centred prescription of physical activity and exercise in addition to standard care.
  Interventions: Other: Physical activity
- Control group (No Intervention): This group will receive standard care.

INTERVENTIONS:
Other: Physical activity — The intervention group will receive an individualized and person-centred prescription of physical activity and exercise.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn about physical activity's effect on health in people who have had surgery of a non-functioning pituitary adenoma.

The main questions it aims to answer are:

* Do physical activity increase quality of life?
* Do physical activity increase general health, cardiovascular fitness, self-efficacy and muscle strength and reduce fatigue and cardiovascular risk profile?

Participants will at the start of the the study, at 6 months follow up and 12 months follow up:

* Fill out health surveys
* Perform a cycling test, hand strength test, chair stand test and wear and accelerometer for a week
* Undergo a dual energy X-ray absorptiometry to measure muscle and fat mass
* Leave blood samples

Researchers will compare those who are randomized to the intervention and see a physiotherapist to get an individualized and person-centred prescription of physical activity plan and those who are randomized not to be in the intervention to see if physical activity increases quality of life and general health.¨.

DETAILED DESCRIPTION:
This study is an unblinded, prospective, randomized, controlled trial where 120 participants will be assigned to either an intervention group or a control group - 60 in each arm. The intervention will receive an individualized and person-centred prescription of physical activity and exercise. The control group will get standard care.

Inclusion criteria

* Patients with non-functioning pituitary adenoma treated with surgery the last ten years
* Stable hormone replacement therapy ≥ 6 months
* Age 18-75 years
* Ability to communicate in Swedish.

Exclusion criteria

* Patients with other pituitary tumours than non-functioning pituitary adenoma
* Patients who could need tumour intervention (surgery or radiotherapy), within one year
* Co-morbidities that could have significant impact on the outcome variables

After the randomization, patients in intervention arm will meet a physiotherapist and a research nurse. The participants will be asked to describe their life situation and experiences regarding their health, diseases, physical activity and exercise and after this be given an individualized and person-centred prescription of physical activity. The exercise will be documented in the self-care plan. In order to assess participants adherence to exercise, participants will be informed to document their performed exercise in the self-care plan during the first 12 weeks. All patients in the intervention group will be followed at 4, 8 and 12 weeks after inclusion in the study when they meet with the same nurse and physiotherapist as at the first visit.

Regarding outcome measures the primary endpoint and the secondary endpoints and will be measured at baseline, and at 6 and 12 months for both the intervention group and the standard care group. The primary endpoint is quality of life and the secondary endpoints are changes in health status, physical activity, cardiorespiratory fitness, muscle strength, self-reported fatigue and self-efficacy, and changes in cardiovascular risk profile.

To assess this the participant will:

* Fill out health surveys
* Perform a cycling test, hand strength test, chair stand test and wear and accelerometer for a week
* Undergo a dual energy X-ray absorptiometry to measure muscle and fat mass
* Leave blood samples

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically significant non-functioning pituitary adenoma treated with surgery during the last ten years
* Stable hormone replacement therapy ≥ 6 months
* Ability to communicate in Swedish.

Exclusion Criteria:

* Patients with any other pituitary tumors than non-functioning pituitary adenoma
* Patients who possibly need tumor intervention, either with surgery or radiotherapy, within one year
* Other diseases or co-morbidities that may have significant impact on the outcome variables, including:
* Ongoing substance abuse and/or untreated psychiatric disorder, including psychoses and bipolar disease (except treatment with SSRI (Selective Serotonin Reuptake Inhibitor) and or SNRI (Serotonin-Norepinephrine Reuptake Inhibitor) for mild/moderate depression and/or anxiety which is allowed).
* Medical therapy with opioids, sedatives or hypnotics (besides treatment with zopiclone and zolpidem which are allowed).
* Current or previous history of neurological diseases with impaired mobility.
* High alcohol consumption (more than 14 alcohol units per week)
* Ongoing treatment for cancer.
* Uncontrolled hypertension or presence of clinically significant cardiac disease
* Severe respiratory insufficiency.
* Severely impaired hepatic function (ALT (Alanine Aminotransferase) and/or AST (Aspartate Aminotransferase) concentrations two times above the upper limit of normal).
* Severely impaired renal function (Glomerular filtration rate <45 ml/min).
* Untreated hypo- or hyperthyroidism
* Pregnancy or breast feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life | At baseline
  Measured with the Short Form Survey Instrument (SF-36), where the score is transformed to a scale 0-100 where 100 represents be best possible health status and quality of life..
Changes in quality of life | At 6 months follow up
  Measured with the Short Form Survey Instrument (SF-36), where the score is transformed to a scale 0-100 where 100 represents be best possible health status and quality of life..
Changes in quality of life | At 12 months follow up
  Measured with the Short Form Survey Instrument (SF-36), where the score is transformed to a scale 0-100 where 100 represents be best possible health status and quality of life..

SECONDARY OUTCOMES:
Changes in health status | At baseline
  Measured with EuroQol-5D (EQ5D). The EuroQol-5D (EQ-5D) index ranges from 0 to 1, where 1 represents the best possible health state, and a visual analog scale (VAS), a scale from 0 to 100, with 100 representing the best imaginable health state.
Changes in health status | At 6 months follow up
  Measured with EuroQol-5D (EQ5D). The EuroQol-5D (EQ-5D) index ranges from 0 to 1, where 1 represents the best possible health state, and a visual analog scale (VAS), a scale from 0 to 100, with 100 representing the best imaginable health state.
Changes in health status | At 12 months follow up
  Measured with EuroQol-5D (EQ5D). The EuroQol-5D (EQ-5D) index ranges from 0 to 1, where 1 represents the best possible health state, and a visual analog scale (VAS), a scale from 0 to 100, with 100 representing the best imaginable health state.
Changes in fitness/muscle strength - Cycling | At baseline
  Cycling test
Changes in fitness/muscle strength - Cycling | At 6 months follow-up
  Cycling test
Changes in fitness/muscle strength - Cycling | At 12 months follow up
  Cycling test
Changes in fitness/muscle strength - Hand strength | At baseline
  Hand strength test
Changes in fitness/muscle strength - Hand strength | At 16 months follow up
  Hand strength test
Changes in fitness/muscle strength - Hand strength | At 12 months follow up
  Hand strength test
Changes in fitness/muscle strength - Chair stand | At baseline
  Chair stand test
Changes in fitness/muscle strength - Chair stand | At 6 months follow up
  Chair stand test
Changes in fitness/muscle strength - Chair stand | At 12 months follow up
  Chair stand test
Changes in fitness/muscle strength - Accelerometer | At baseline
  Accelerometer for a week
Changes in fitness/muscle strength - Accelerometer | At 6 months follow up
  Accelerometer for a week
Changes in fitness/muscle strength - Accelerometer | At 12 months follow up
  Accelerometer for a week
Changes in self-reported self-efficacy | At baseline
  Self-reported self-efficacy through Self-Efficacy t Manage Chronic Disease (a questionnaire with 6 question where you rate yourself 1-10)
Changes in self-reported self-efficacy | At 6 months follow up
  Self-reported self-efficacy through Self-Efficacy t Manage Chronic Disease (a questionnaire with 6 question where you rate yourself 1-10)
Changes in self-reported self-efficacy | At 12 months follow up
  Self-reported self-efficacy through Self-Efficacy t Manage Chronic Disease (a questionnaire with 6 question where you rate yourself 1-10)
Changes in cardiovascular risk profile - Blood pressure | At baseline
  Blood pressure - systolic and diastolic
Changes in cardiovascular risk profile - Blood pressure | At 6 months follow up
  Blood pressure - systolic and diastolic
Changes in cardiovascular risk profile - Blood pressure | At 12 months follow up
  Blood pressure - systolic and diastolic
Changes in cardiovascular risk profile - Blood samples | At baseline
  Blood lipids
Changes in cardiovascular risk profile - Blood samples | At 6 months follow up
  Blood lipids
Changes in cardiovascular risk profile - Blood samples | At 12 months follow up
  Blood lipids

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Univesity Hospital, Gothenburg, Västra Götaland County, Sweden